CLINICAL TRIAL: NCT06074432
Title: Risk Factors Associated With Morbidity and Mortality in Emergency Colorectal Cancer Resections
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Turgut Donmez, Associate Professor, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: Emer. CRC Mort Risk Factors
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
Keywords: Emergency Treatment; Colorectal Cancer; Mortality; Morbidity; Risk Factors
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency Colorectal Cancer Resection: Patients that underwent emergent resection because of histopathologically confirmed colorectal carcinoma
  Interventions: Other: Emergency Colorectal Resection

INTERVENTIONS:
Other: Emergency Colorectal Resection — Patients underwent resection due to colorectal carcinoma in emergency surgery

SUMMARY:
Study is designed to investigate the risk factors associated with morbidity and mortality in patients who underwent emergency resection because of colorectal cancer in general surgery clinic of a tertiary referral hospital.

DETAILED DESCRIPTION:
Patients who underwent emergency colorectal resection in a single tertiary referral center between January 2019 and December 2022 were planned to include. All patients were equal or older than 18 years and histopathologically found to have primary colorectal malignant neoplasms.

Patients were excluded from the analysis if they met any of the following criteria: patients underwent surgery without resection, patients operated with a different indication from primary colorectal cancer such as diverticulitis, ischemia, inflammatory bowel diseases or metastases of another malignancy. Patients with insufficient clinical data were also excluded.

Surgical procedures were performed by general surgeons and only some of them had a subspecialisation in colorectal surgery.

Factors such as age, sex, body mass index (BMI), ASA score, Charlson comorbidity index, smoking status and comorbidity histories, existence of perioperative blood transfusions, duration of surgery, length of hospital stay, tumor side and characteristics, presence of perforation and ascites of the cases were noted. Patients were divided into two subgroups in terms of ASA scores. ASA I and II patients were the first subgroup and ASA III and IV were the other subgroup. A tumor located distal to the midpoint of the transverse colon was accepted as left sided and the others as proximal right sided.

Nutritional risk screening (NRS 2002) scores of the patients were also included in the analyzes. NRS 2002 scores were recorded at hospital admission. Patients were divided into two subgroups as being at nutritional risk (score 3 or more) or not (score less than 3) according to the total score recorded. For the presence of morbidity, a Clavien-Dindo score of 3 and more complications were taken as basis. Mortality was defined as the death within 90 days of operation.

Risk factors for both morbidity and mortality were first evaluated using univariate analyzes. Factors detected as significantly related to morbidity and mortality in appropriate univariate analyzes were included in multivariate analyzes with logistic regression. Multivariate analyzes done for both morbidity and mortality. The effects of risk factors on morbidity and mortality were expressed as the relative risk (odds ratio) with their 95% confidence intervals. Statistical significance level was set at 0.05

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent emergency colorectal resection between January,1 2019 and December,31 2022 were included. All patients were equal or older than 18 years and histopathologically found to have primary colorectal malignant neoplasms

Exclusion Criteria:

* Patients operated with a different indication from primary colorectal cancer such as diverticulitis, ischemia, inflammatory bowel diseases or metastases of another malignancy
* Patients with insufficient clinical data were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent emergency colorectal resection between January 2019 and December 2022
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Morbidity | Until postoperative 90 days
  Patients developed a major complication that has a Clavien-Dindo Score ≥3
Mortality | Until postoperative 90 days
  Patients died in the postoperative period within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Karabulut, Study Chair — University of Health Sciences, Bakirkoy Dr.Sadi Konuk Training and Research
Locations (1):
- Bakırkoy Dr.Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No